CLINICAL TRIAL: NCT06039592
Title: A Prospective Controlled Study for the Treatment Effect of Different Intervention Strategies for Pediatric Mitral Regurgitation--A Multicenter Prospective Cohort Study of Innovative Drug Therapy in Improving Left Ventricular Function After Mitral Repair
Brief Title: Study of Innovative Drug Strategies in Improving Left Ventricular Function After Mitral Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Shanghai Children's Medical Center (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Shoujun Li, Director of Congenital Heart Surgery Center, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-GSP-GG-19-3
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Congenital Mitral Insufficiency
Keywords: congenital heart disease; mitral regurgitation; mitral valve repair postoperative; drug therapy
MeSH Terms: conditions — Heart Defects, Congenital; Mitral Valve Insufficiency | interventions — Captopril; Metoprolol; Spironolactone; Torsemide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Modified Drug Therapy Group: Patient in this group will undergo a one-year course of medication, including Captopril(tablet, 0.3mg/kg, tid), Metoprolol(tablet, 0.2mg/kg, bid), Spironolactone(tablet, 2-4mg/kg, bid), Torsemide(tablet, 0.2-0.5mg/ mg, bid), and Potassium Citrate(powder, 0.06g/kg, tid).
  Interventions: Drug: Captopril Tablets; Drug: Metoprolol Oral Tablet; Drug: Spironolactone Tablets; Drug: Torsemide Tablets; Drug: Potassium citrate powder
- Traditional Drug Therapy Group: Patient in this group will undergo a one-year course of medication, including Torsemide(tablet, 0.2-0.5mg/mg, bid) and Potassium Citrate(powder, 0.06g/kg, tid).
  Interventions: Drug: Torsemide Tablets; Drug: Potassium citrate powder

INTERVENTIONS:
Drug: Captopril Tablets — 0.3mg/kg, tid
  Groups: Modified Drug Therapy Group
Drug: Metoprolol Oral Tablet — 0.2mg/kg, bid
  Groups: Modified Drug Therapy Group
Drug: Spironolactone Tablets — 2-4mg/kg, bid
  Groups: Modified Drug Therapy Group
Drug: Torsemide Tablets — 0.2-0.5mg/mg, bid
Drug: Potassium citrate powder — 0.06g/kg, tid

SUMMARY:
The goal of this observational study is to compare the safety and effectiveness of a modified drug therapy with traditional drug therapy in pediatric patients after mitral repair.

The main questions it aims to answer are:

* Can a modified drug therapy improve both left ventricular and mitral valve function in pediatric patients after mitral repair?
* Can the adverse drug reactions caused by the modified drug therapy be non-inferior (clinically acceptable) to those of the traditional drug therapy? Participants will be assigned to either the Modified Drug Therapy Group (comprising angiotensin-converting enzyme inhibitor (ACE-I), beta-blockers, diuretics, potassium supplements, and spironolactone) or the Traditional Drug Therapy Group (diuretics and potassium supplements) based on personal preferences and clinical assessments by their attending physicians. They will undergo a 6-months course of medication. Additionally, echocardiography, electrocardiograms, complete blood counts, biochemical tests, and measurements of N-terminal pro-brain natriuretic peptide (NT-proBNP) were conducted before the initiation of medication therapy and at 1 month, 3 months, and 6 months after treatment commencement. Researchers will compare the Modified Drug Therapy Group and the Traditional Drug Therapy Group to see if the recurrence rate of moderate to severe mitral valve regurgitation, as assessed by echocardiography after 6 months of treatment, is lower in the former than in the latter.

ELIGIBILITY:
Inclusion Criteria:

* under 14 years old
* after mitral valve repair

Exclusion Criteria:

* Patients with heart failure requiring ventricular assist or cardiac synchronization therapy
* Patients with severe pulmonary hypertension (pulmonary arterial pressure >6 Wood·U)
* Patients with severe liver and kidney failure
* Patients who are allergic to related medications
* Patients with symptomatic hypotension who cannot tolerate related drugs

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of 14 after mitral valve repair surgery.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of moderate to severe mitral valve regurgitation | after 12 months of treatment
  During follow-up visits, echocardiographic examination is conducted to measure the degree of mitral valve regurgitation. If it falls within the moderate to severe range, it is recorded as a recurrence.

SECONDARY OUTCOMES:
Improvement in symptoms | after 12 months of treatment
  Based on patient and caregiver descriptions, if symptoms such as chest discomfort, shortness of breath, and delayed development show improvement following physical activity, it is recorded as an improvement in symptoms.
Improvement in left ventricular function | after 12 months of treatment
  Based on the echocardiogram, measurements are taken for left ventricular ejection fraction, left ventricular fractional shortening, left ventricular end-diastolic diameter, left ventricular end-diastolic volume, left ventricular end-systolic diameter, and left ventricular end-systolic volume.
NT-proBNP level | after 12 months of treatment
  The trend in NT-proBNP levels.
Incidence rate of drug adverse reactions | after 12 months of treatment
  The incidence of abnormalities in complete blood count, electrolytes, liver and kidney function, and cardiac enzymes.

CONTACTS AND LOCATIONS:
Overall Officials: Shoujun Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No